CLINICAL TRIAL: NCT01145326
Title: Functional Microarray Augmentation of Skin Treatment With Lidocaine (FAST Lidocaine)
Brief Title: Functional Microarray Augmentation of Skin Treatment With Lidocaine
Acronym: FAST
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The device is undergoing further study in China, per FDA requirements.
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OUDEM 2010-1
Record Dates: First submitted 2010-06-14; First posted 2010-06-16 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Pain Perception; Phlebotomy
Keywords: venipuncture; phlebotomy; pain perception

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Sham Comparator): Sham-Functional microneedles (no actual microneedles) application, prior to 4% lidocaine gel (LG4) placement.
  Interventions: Drug: 4% lidocaine gel application with sham microneedle device
- Microneedle (Experimental): Functional microarray (FMA) (microneedles) application, prior to 4% lidocaine gel (LG4) placement.
  Interventions: Drug: Microneedle-facilitated lidocaine application

INTERVENTIONS:
Drug: 4% lidocaine gel application with sham microneedle device — Topical 4% lidocaine gel (LG4) applied to subject, after application of sham microneedle device (FMA).
  Other Names: 4% Lidocaine gel with sham-functional microarray (FMA)
  Arms: Control
Drug: Microneedle-facilitated lidocaine application — Application of 4% lidocaine gel (LG4), after application of microneedle (FMA) device
  Other Names: 4% lidocaine gel with functional microarray
  Arms: Microneedle

SUMMARY:
The purpose of this study is to determine whether co-application of a functional microarray of needles (FMA) speeds the rate at which topical anesthesia is provided. A secondary goal is to determine whether the depth of anesthesia is enhanced.

DETAILED DESCRIPTION:
The study's primary goal is to determine whether co-application of a functional microarray of needles (FMA) speeds the rate at which topical anesthesia is provided by lidocaine gel 4% (LG4). A secondary goal is to determine whether the depth of anesthesia is enhanced.

ELIGIBILITY:
Inclusion Criteria: age at least 18 years, must provide voluntary consent, weight at least 50 kg, no allergies to lidocaine, no skin disease, inflammation, or infection at the venipuncture sites to be tested

Exclusion Criteria: cannot have any major dermatologic disease history, known liver abnormalities, women who are currently breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Venipuncture pain levels | 1 hour

SECONDARY OUTCOMES:
Undesirable side effects | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Stephen H. Thomas, MD MPH, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Schusterman Clinic, Tulsa, Oklahoma, United States